CLINICAL TRIAL: NCT02349867
Title: A Phase 1 Study of Neoadjuvant Chemotherapy, Followed by Concurrent Chemoradiation With Gemcitabine, Sorafenib, and Vorinostat in Pancreatic Cancer
Brief Title: Neoadjuvant Chemotherapy Followed by Radiation Therapy and Gemcitabine/Sorafenib/Vorinostat in Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12-07328; NCI-2015-00017 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC-12-07328 (Other: Virginia Commonwealth University/Massey Cancer Center); P30CA016059 (NIH)
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Pancreatic Adenocarcinoma; Stage IA Pancreatic Cancer; Stage IB Pancreatic Cancer; Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer; Recurrent Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Sorafenib; Vorinostat; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (chemotherapy, chemoradiation) (Experimental): Participants receive gemcitabine IV infusion over 30 minutes (200 mg/m2 weekly) x 6, concurrent administration of oral sorafenib and oral vorinostat (both per dose-escalation schema), and concurrent RT( 3-Dimensional Conformal Radiation Therapy or Intensity-Modulated Radiation Therapy) administered at 1.8-Gy fractions to a total dose of 50.4 Gy over 5 ½ weeks (28 daily fractions).
  Interventions: Drug: Gemcitabine; Drug: Sorafenib; Drug: Vorinostat; Radiation: 3-Dimensional Conformal Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Other: RosetteSep; Other: DEPfff

INTERVENTIONS:
Drug: Gemcitabine — Given IV
  Other Names: dFdC; dFdCyd
Drug: Sorafenib — Given PO
  Other Names: BAY 54-9085; Nexavar; SFN
Drug: Vorinostat — Given PO
  Other Names: L-001079038; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3D CRT
  Other Names: 3D-CRT; Conformal Therapy; Radiation Conformal Therapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy
Other: RosetteSep — Circulating tumor cells (CTCs) will be captured and analyzed, when detected. Pancreatic cancer has been a difficult tumor in which to detect CTCs (41). Utilization of techniques that do not require cell surface marker expression will be explored. Samples will either be analyzed by negative-selection techniques (RosetteSep). Peripheral blood samples will be collected at several time-points for CTC enumeration and to evaluate CD95 density.
  Other Names: negative-selection techniques
Other: DEPfff — Circulating tumor cells (CTCs) will be captured and analyzed, when detected. Pancreatic cancer has been a difficult tumor in which to detect CTCs (41). Utilization of techniques that do not require cell surface marker expression will be explored. Samples will either be analyzed by with the ApoStream dielectrophoretic field-flow fractionation (DEPfff) enrichment device. Peripheral blood samples will be collected at several time-points for CTC enumeration and to evaluate CD95 density.
  Other Names: ApoStream dielectrophoretic field-flow fractionation

SUMMARY:
Determine the doses and schedule appropriate for phase 2 study of sorafenib and vorinostat with concurrent gemcitabine and radiation therapy (RT) as neoadjuvant treatment of pancreatic cancer following chemotherapy. Recommended phase II dose RP2Ds and schedule of sorafenib and vorinostat defined as the doses and schedule that are the same as or less than the maximum tolerated dose (MTD) and schedule.

DETAILED DESCRIPTION:
This is a phase 1 study of concurrent chemoradiation using a regimen of sorafenib and vorinostat with gemcitabine and radiation following chemotherapy in patients with pancreatic cancer to find the recommended phase II dose (RP2D) of the concurrent chemoradiation combination. A traditional 3+3 dose-escalation design will be conducted for the sorafenib and vorinostat dose escalation. Adenocarcinoma of the pancreas without distant metastasis that has been treated with ≥ 1 prior therapy (not including radiation) encompassing at least 2 months. Adequate hematologic, hepatic, and renal function. Ability to take oral medication. To determine the doses and schedule appropriate for phase 2 study of sorafenib and vorinostat with concurrent gemcitabine and radiation therapy (RT) as neoadjuvant treatment of pancreatic cancer following chemotherapy.This is a dose-escalation trial employing a standard "3+3" schema of sorafenib and vorinostat.

ELIGIBILITY:
Inclusion Criteria:

* Adenocarcinoma of the pancreas
* Prior therapy with ≥ 1 prior systemic therapy over a period of at least 2 months (eg, at least two 4-week cycles of a regimen such as gemcitabine and nab-paclitaxel; or at least four 2-week cycles of a regimen such as FOLFOX, FOLFIRINOX, or FOLFIRI) -Candidate for additional therapy consisting of radiation with gemcitabine- radiosensitization.
* Able to initiate study treatment no later than 9 weeks from last dose of any antineoplastic component of prior therapy regimen.
* Recovery from ≥ grade 2 toxicities of prior therapy regimen to grade 1 or baseline, with the exception of anemia and lymphopenia and chronic residual toxicities that in the opinion of the investigator are not clinically relevant given the known safety/toxicity profiles of gemicitabine, sorafenib, and vorinostat (eg, alopecia, changes in pigmentation, stable endocrinopathies). Patients with ≤ grade 2 peripheral sensory or motor neuropathy are eligible..
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3 x upper limit of normal (ULN) for the laboratory
* Total bilirubin <= 1.5 x ULN for the laboratory at the time of enrollment, all forms of biliary stents allowed
* Creatinine clearance >= 45 mL/min as calculated by the standard Cockcroft-Gault equation using age, actual weight, creatinine and gender
* International normalized ratio (INR) <= 1.5
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3 (may not be transfused to meet this level for enrollment)
* Measurable or evaluable disease by Response Evaluation Criteria in Solid Tumors (RECIST) (version [v]1.1
* Ability to understand and the willingness to sign a written informed consent document
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use a medically accepted form of birth control during the treatment and for 2 months following completion of study treatment

Exclusion Criteria:

* Prior radiotherapy for pancreatic cancer
* Prior surgical resection of pancreatic cancer
* Evidence of metastatic disease
* Any investigational agent within 4 weeks of study treatment initiation
* Diagnosis or treatment for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, any in situ malignancy, or low-risk prostate cancer after curative therapy
* Intolerance of protocol agents as follows:

  * Known or presumed intolerance of gemcitabine, vorinostat or sorafenib
  * Experienced any of the following toxicities with prior gemcitabine adminstration (if given): capillary leak syndrome, posterior reversible encephalopathy, hemolytic uremic syndrome, thrombotic thrombocytopenic purpura, unexplained dyspnea or other evidence of severe pulmonary toxicity, or severe hepatic toxicity
* Unable to swallow medication
* Suspected malabsorption or obstruction; note: use of pancreatic enzyme supplements is allowed to control malabsorption
* Contraindication to antiangiogenic agents, including:

  * Bronchopulmonary hemorrhage/bleeding event >= grade 2 (Common Terminology Criteria for Adverse Events [CTCAE] v4.0) within 12 weeks prior to of treatment
  * Any other hemorrhage/bleeding event >= grade 3 (CTCAE v4.0) within 12 weeks prior to initiation of treatment
  * Serious non-healing wound, ulcer, or bone fracture
* Arterial thrombotic or embolic events such as a myocardial infarction or cerebrovascular accident (including transient ischemic attacks) within the 6 months prior to initiation of treatment. Incidental clinically insignificant embolic phenomena that do not require anti-coagulants are not excluded. Also,tumor-associated thrombus of locally-involved vessels does not count as an exclusion criterion.
* Clinically significant cardiac disease, including major cardiac dysfunction, such as uncontrolled angina, clinical congestive heart failure with New York Heart Association (NYHA) class III or IV, ventricular arrhythmias requiring anti-arrhythmic therapy, recent (within 6 months) myocardial infarction or unstable coronary artery disease
* Concomitant use of other histone deacetylase (HDAC) inhibitors
* Planned ongoing administration of STRONG cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducers. Examples of clinical inducers and classifications of strong, moderate, and weak interactions are available through the FDA website (Table 3-3 of website): http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm
* Persistent heart rate (HR) < 50 or > 120 beats per minute (bpm).
* QT(c) ≥ 481 ms (>= grade 2) on electrocardiogram (ECG) prior to initiation of treatment

  * If baseline QTc on screening ECG meets exclusion criteria:

    * Check potassium and magnesium serum levels
    * Correct any identified hypokalemia and/or hypomagnesemia and repeat ECG to confirm exclusion of patient due to QTc
  * For patients with HR >60 of >100 beats per minute (bpm), no manual read of QTc is required
  * For patients with baseline HR < 60 or > 100 bpm, manual read of QT by cardiologist is required, with Fridericia correction applied to determine QTc
* Planned ongoing treatment with other drugs thought to potentially adversely interact with study drugs; if such medications have been used, patients must be off of these agents for >= 2 weeks prior to initiation of treatment:

  * Anticoagulants at therapeutic doses
  * Immunosuppressants such as tacrolimus, leflunomide or tofacitinib, roflumilast, pimecrolimus
* Serious uncontrolled infection > grade 2 (CTCAE v4.0)
* Medical, psychological, or social conditions that, in the opinion of the investigator, may increase the patient's risk or interfere with the patient's participation in the study or hinder evaluation of the study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01-29 (Actual); Primary Completion 2020-05-13 (Actual); Study Completion 2022-05-13 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose and schedule | 18-36 months
  Determine the doses and schedule appropriate for phase 2 study of sorafenib and vorinostat with concurrent gemcitabine and radiation therapy (RT) as neoadjuvant treatment of pancreatic cancer following chemotherapy.

SECONDARY OUTCOMES:
Number of participants with adverse events using National Cancer Institute CTCAE v4.0 | Up to 30 days following last administration of the chemoradiation treatment
  Adverse events using NCI Common Terminology Criteria for Adverse Events, Version 4.0. Adverse events will be listed and summary descriptive statistics will be calculated.
Tumor response (complete response or partial response) measured using RECIST version 1.1 | Up to 2 years
  Evaluate number of participants with tumor response measured using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. At the completion of concurrent chemoradiation. Tumor response will be measured as complete response, partial response, stable disease, or tumor progression.
Surgery | Up to 2 years
  Number of participants able to undergo resection after neoadjuvant therapy (chemotherapy followed by concurrent chemoradiation)
R0 Resection rate | Up to 2 years
  Determine the number of patients able to undergo margin-negative resection following neoadjuvant therapy.
Progression-free survival (PFS) | Up to 2 Years
  Number of participants with progression free survival (PFS) defined as the percentage of patients able to undergo margin-negative resection following neoadjuvant therapy
Overall Survival | Up to 2 Years
  The number of participants with overall survival (OS) defined as the time from the date of diagnosis until death by any cause

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia, United States

REFERENCES:
- [Derived] Booth L, Poklepovic A, Dent P. Neratinib decreases pro-survival responses of [sorafenib + vorinostat] in pancreatic cancer. Biochem Pharmacol. 2020 Aug;178:114067. doi: 10.1016/j.bcp.2020.114067. Epub 2020 Jun 3. PMID 32504550